CLINICAL TRIAL: NCT05039047
Title: External Validation of Two Prediction Models for Independent Gait After Stroke
Acronym: REPEAT
Status: Terminated | Type: Observational
Why Stopped: Change position of PI, no replacement available, therefore unable to continue recruitment - all enrolled patients finished the study according to plan
Sponsor: Janne Veerbeek (Other)
Responsible Party: Sponsor-Investigator, Janne Veerbeek, PT, PhD, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Other Study IDs: BASEC-ID 2021-01519
Record Dates: First submitted 2021-08-18; First posted 2021-09-09 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Gait; Prognosis; External validation; EPOS model; TWIST model; Falls
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort
  Interventions: Other: Standard stroke acute care and rehabilitation

INTERVENTIONS:
Other: Standard stroke acute care and rehabilitation — According to Swiss national guidelines and local protocols

SUMMARY:
Regaining independent gait is one of the main goals in stroke rehabilitation and early prediction of gait outcome is important to guide discharge planning at acute stroke units, design rehabilitation and inform patients and relatives. In the last decade, two easy-to-apply prediction models for gait were developed: the EPOS model in the Netherlands and the TWIST model in New Zealand. Although the models' performance in the development cohorts was good, this does not automatically mean that the models are ready for application in clinical practice, as it is unknown whether their performance is also good in an independent cohort from a different country and with different patient characteristics. Such external validation is an essential step towards clinical implementation of prediction models.

A mobility-related problem is the occurrence of falls after stroke. Walking is among the Top 3 activities during which stroke patients fall, with the other two activities being transferring or sitting in a wheelchair. Especially soft tissue injuries after a fall are common and in 1-15% of the patients, the fall results in a fracture. Apart from the costs that arise from these injuries, falls have a negative impact on the patient's physical functioning and psychological status, with an increased dependency and fear of falling, resulting in a reduced quality of life.

A systematic review found 12 studies that developed fall risk prediction models for either inpatient rehabilitation stroke patients or those living in the community. Important predictors for falls are the presence of hemi-inattention, fall history and balance deficits. However, none of the models had an acceptable performance and predictors were not always captured by a validated assessment, which is an important prerequisite for an unbiased prediction model.

The primary aim of this study is to externally validate the EPOS and TWIST models for independent gait after stroke in a heterogeneous sample of subjects admitted to the hospital with an acute stroke. It is hypothesized that the performance of both models in this independent cohort will be lower than in the development cohorts, but still be adequate.

The secondary objective is to investigate the occurrence and predictability of falls within the first six months after stroke and its relationship with the prognosis for independent gait within this sample.

ELIGIBILITY:
Inclusion criteria:

* First-ever or recurrent stroke as confirmed by computerized tomography and/ or magnetic resonance imaging
* Not able to walk independently within the first 72 hours after stroke (Functional Ambulation Categories <4)
* Age ≥18 year
* Written informed consent

Exclusion criterion:

• Not able to walk independently before hospital admission (Functional Ambulation Categories <4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to a hospital with an acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories (0-5 points, higher scores being better) | 6 weeks poststroke
  Walking ability (independence)
Functional Ambulation Categories (0-5 points, higher scores being better) | 12 weeks poststroke
  Walking ability (independence)
Functional Ambulation Categories (0-5 points, higher scores being better) | 26 weeks poststroke
  Walking ability (independence)

SECONDARY OUTCOMES:
Falls | 6 weeks poststroke
  Number of falls
Falls | 12 weeks poststroke
  Number of falls
Falls | 26 weeks poststroke
  Number of falls

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (0-42 points, lower scores being better) | Hospital admission, usually within 24 hours poststroke
  Neurological functions
Trunk Control Test (0-100 points, higher scores being better) | within 72 hours poststroke
  Trunk control
Motricity Index - lower extremity subscale (0-100 points, higher scores being better) | within 72 hours poststroke
  Lower extremity isometric muscle strength
Medical Research Grading - hip extension (0-5 points, higher scores being better) | within 72 hours poststroke
  Hip extension muscle strength
Modified Rankin Scale (0-5 points, lower scores being better) | 6 weeks poststroke
  Global disability
Modified Rankin Scale (0-5 points, lower scores being better) | 12 weeks poststroke
  Global disability
Modified Rankin Scale (0-5 points, lower scores being better) | 26 weeks poststroke
  Global disability

CONTACTS AND LOCATIONS:
Overall Officials: Janne M. Veerbeek, PhD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veerbeek JM, Van Wegen EE, Harmeling-Van der Wel BC, Kwakkel G; EPOS Investigators. Is accurate prediction of gait in nonambulatory stroke patients possible within 72 hours poststroke? The EPOS study. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):268-74. doi: 10.1177/1545968310384271. Epub 2010 Dec 26. PMID 21186329
- [Background] Smith MC, Barber PA, Stinear CM. The TWIST Algorithm Predicts Time to Walking Independently After Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):955-964. doi: 10.1177/1545968317736820. Epub 2017 Nov 1. PMID 29090654
- [Background] Steyerberg EW, Moons KG, van der Windt DA, Hayden JA, Perel P, Schroter S, Riley RD, Hemingway H, Altman DG; PROGRESS Group. Prognosis Research Strategy (PROGRESS) 3: prognostic model research. PLoS Med. 2013;10(2):e1001381. doi: 10.1371/journal.pmed.1001381. Epub 2013 Feb 5. PMID 23393430
- [Background] Moons KGM, Wolff RF, Riley RD, Whiting PF, Westwood M, Collins GS, Reitsma JB, Kleijnen J, Mallett S. PROBAST: A Tool to Assess Risk of Bias and Applicability of Prediction Model Studies: Explanation and Elaboration. Ann Intern Med. 2019 Jan 1;170(1):W1-W33. doi: 10.7326/M18-1377. PMID 30596876
- [Background] Moons KG, Kengne AP, Grobbee DE, Royston P, Vergouwe Y, Altman DG, Woodward M. Risk prediction models: II. External validation, model updating, and impact assessment. Heart. 2012 May;98(9):691-8. doi: 10.1136/heartjnl-2011-301247. Epub 2012 Mar 7. PMID 22397946
- [Background] Lamb SE, Jorstad-Stein EC, Hauer K, Becker C; Prevention of Falls Network Europe and Outcomes Consensus Group. Development of a common outcome data set for fall injury prevention trials: the Prevention of Falls Network Europe consensus. J Am Geriatr Soc. 2005 Sep;53(9):1618-22. doi: 10.1111/j.1532-5415.2005.53455.x. PMID 16137297
- [Background] Batchelor FA, Mackintosh SF, Said CM, Hill KD. Falls after stroke. Int J Stroke. 2012 Aug;7(6):482-90. doi: 10.1111/j.1747-4949.2012.00796.x. Epub 2012 Apr 12. PMID 22494388
- [Background] Walsh M, Galvin R, Horgan NF. Fall-related experiences of stroke survivors: a meta-ethnography. Disabil Rehabil. 2017 Apr;39(7):631-640. doi: 10.3109/09638288.2016.1160445. Epub 2016 Mar 23. PMID 27008035
- [Background] Walsh ME, Galvin R, Boland F, Williams D, Harbison JA, Murphy S, Collins R, Crowe M, McCabe DJH, Horgan F. Validation of two risk-prediction models for recurrent falls in the first year after stroke: a prospective cohort study. Age Ageing. 2017 Jul 1;46(4):642-648. doi: 10.1093/ageing/afw255. PMID 28104593